CLINICAL TRIAL: NCT02109601
Title: Tablet Computers for Hospitalized Adults: a Novel Approach to Increasing Patient Engagement With Their Electronic Personal Health Records
Brief Title: Patient-Centered Tablets: Applications for Inpatient Admissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-09854
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Mobile Health
Keywords: Patient Portals; Personal Health Records; Patient Engagement; Mobile Health; Tablet Computers
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control patients receive iPad tablets during their hospital stay with only LIMITED bedside training from a research assistant on how to access and effectively use their patient portal.
  Interventions: Other: Limited bedside training on patient portal use.
- Intervention (Experimental): Intervention patient receive iPad tablets during their hospital stay with EXTENSIVE bedside training from a research assistant on how to access and effectively use their patient portal.
  Interventions: Other: Extensive bedside training for accessing patient portal

INTERVENTIONS:
Other: Extensive bedside training for accessing patient portal — EXTENSIVE bedside training from a research assistant on how to access and effectively use their patient portal.
  Other Names: Apple iPad tablets; Epic MyChart patient portal
  Arms: Intervention
Other: Limited bedside training on patient portal use. — EXTENSIVE bedside training from a research assistant on how to access and effectively use their patient portal.
  Arms: Control

SUMMARY:
RESEARCH QUESTION:

Are hospitalized patients able to use a tablet computer (iPad) to take brief surveys, access their patient portal (MyChart), and watch informational videos about their condition?

DETAILED DESCRIPTION:
STUDY DESIGN:

Small pilot study evaluating pre/post impressions of information technology and the feasibility of using a tablet computer for education purposes and to complete a daily survey about preparations for discharge and post-acute care.

The study has two distinct parts. Patients will have the option to participate in either one or both parts.

PART 1: Using iPads to learn about health conditions We will enroll and randomize patients to intervention or control groups. Allocation to be intervention or control group will be determined using a computer-based random number generator. All patients will be orientated to using an iPad, asked to take a pre-use survey, will have a MyChart account set up and view EMMI modules. Intervention group patients will receive specific detailed education about how to access, navigate and use MyChart using tablets (iPads) . Control group patients will not receive this specific education about how to access, navigate and use MyChart using tablets (iPads). Both intervention and control group patients will be asked to complete a post-use survey. We will access MyChart data repositories to determine if patients continue to access their patient portal for up to 30 days after the completion of this part of the study.

PART 2: Using iPads to prepare for discharge We will enrol all eligible patients (regardless of intervention or control group status in Part 1) to complete a daily Readiness for Discharge Survey (RDS). This standardized validated survey will determine a range of discharge and post-acute issues and will be fed back to the patient's health care team. Patient demographic and clinical information will be abstracted from their medical record to determine if there are any specific issues related to specific groups of patients. Initially the RDS will be completed on a paper survey but will be eventually be administered via an iPad.

ELIGIBILITY:
Inclusion Criteria:

Adult patients admitted to any service at UCSF Medical Center

Exclusion Criteria:

Patients not speaking English. Patients unable to give consent. Patients unable to safely use a tablet computer for any reason. Patients being discharged on day of approach. Patient cognitively impaired and unable to give consent. Patient in ICU. Patient in some form of droplet isolation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patient Portal Usage | During and after hospitalization (up to 30 days)
  Effects of iPad intervention to improve patient access to their patient portal will be assessed during hospitalization and for 30 days after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Medical Center (Moffitt-Long Hospital), San Francisco, California, United States

REFERENCES:
- [Derived] Greysen SR, Magan Mendoza Y, Rosenthal J, Jacolbia R, Rajkomar A, Lee H, Auerbach A. Using Tablet Computers to Increase Patient Engagement With Electronic Personal Health Records: Protocol For a Prospective, Randomized Interventional Study. JMIR Res Protoc. 2016 Sep 6;5(3):e176. doi: 10.2196/resprot.4672. PMID 27599452